CLINICAL TRIAL: NCT03367312
Title: Assessing Response to Inhaled Prostacyclin With Hyperpolarized Xe MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor, Duke University Medical Center, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00086282
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Vascular Disease

STUDY DESIGN:
Intervention Model Description: This will be a single-blinded open-label study enrolling 15 patients (accrued 12 subjects total) with Pulmonary Hypertension who are currently on a stable dose of Inhaled Prostacyclin for treatment of PH.
Masking Description: The outcomes assessor, the radiologist who is reading the imaging will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pulmonary Hypertension Patients on Inhaled Prostacyclin (Experimental): 10 subjects will Pulmonary Hypertension on a stable dose of Inhaled Prostacyclin for treatment of PH.
  Interventions: Drug: Hyperpolarized 129Xenon gas

INTERVENTIONS:
Drug: Hyperpolarized 129Xenon gas — Hyperpolarized 129Xenon gas XeMRI scans will provide 3D images of ventilation and gas exchange pre, post, and 2-4 hours post inhaled prostacyclin treatment. Subjects will inhale HP 129Xe from the dose delivery bags with each scan and then move into the scanner and undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will undergo several MRI scans after inhalation of HPXe. This will occur as three scans at the three different time points (pre, post, and 2-4 hours post) of inhaled prostacyclin treatment.
  Other Names: Xe MRI

SUMMARY:
This study seeks to deploy several forms of 129Xe MRI contrast as well as emerging conventional proton MRI techniques for imaging lung structure and perfusion. Specifically, the 129Xe MRI scans will provide 3D images of ventilation and gas exchange, and spectroscopic indices will be evaluated too test gas exchange dynamics with high temporal resolution. The conventional 1H MRi scans will include a free-breathing ultra-short echo time scan that provides images similar to that of a CT scan. This will be done pre, immediately post, and 2-4 hours post inhaled prostacyclin therapy.

DETAILED DESCRIPTION:
This study seeks to determine whether hyperpolarized 129Xenon MRI can detect improvements in pulmonary gas exchange in patients with Group 1 and 3 PH treated with iTRE. We will associate this with changes in serum concentrations of treprostinil and levels of peripheral vasodilation. This work seeks to apply and test a novel non-invasive methodology, hyperpolarized (HP) 129Xenon (Xe) magnetic resonance imaging (MRI), for the diagnosis of Pulmonary Vascular Disease. Hyperpolarized 129Xe MRI has been under active development and used in clinical research at Duke for over 7 years. If successful, 129Xe MRI could overcome the current limitations of PVD diagnosis while conferring a number of potential benefits. First, imaging the abnormalities in the lungs allows the diagnosis of PVD in the setting of concomitant heart or lung disease. With HP 129Xe MRI, abnormalities in gas exchange secondary to PVD can be directly visualized. Second, non-invasive diagnosis of PVD could remove the need for an invasive RHC. While RHC is a relatively safe procedure, there are a number of limitations to the interpretation of RHC, including arbitrary cutoffs for mPAP, PCWP, and PVR. Third, the abnormalities on HP 129Xe MRI could be used to non-invasively monitor response to therapy. If we are successful in demonstrating the applicability of HP 129Xe MRI, this technology holds the promise of greatly improving the diagnosis and management of PVD.

This study will enroll ten patients with pulmonary hypertension (PH). The ten patients will be World Health Organization (WHO) PH classification Group 1 or out-of-proportion Group 3, with lung disease. These patient have been inhaled treprostinil (iTRE) as standard of care for their PH. Inhaled treprostinil (iTRE) is an FDA approved medication under the brand name of Tyvaso. The major pharmacologic actions of treprostinil are direct vasodilation of pulmonary and systemic arterial vascular beds and inhibition of platelet aggregation. The medication is delivered noninvasively, directly to the lungs using the approved ultrasonic nebulizer delivery system. Patients will take the inhaled treatment four times a day, about every four hours.

The iTRE will be used to characterize their 129Xe MRI imaging, peripheral vasodilation and serum treprostinil concentration before and after treatment with iTRE. As iTRE has a plasma concentration half-life of ~ 45 minutes and time-to-peak concentration of 15 minutes, imaging done immediately before, 15 minutes after and 2-4 hours after drug treatment would potentially allow the visualization of changes in gas diffusion and peripheral vasodilation associated with iTRE. This is similar to changes seen in changes in ventilation in asthma after treatment with bronchodilators. Monitoring a later time point would also allow us to test whether vasodilation persists in the lung vasculature compared to the peripheral circulation. This study seeks to deploy several forms of 129Xe MRI contrast as well as emerging conventional proton MRI techniques for imaging lung structure and perfusion. Specifically, the 129Xe MRI scans will provide 3D images of ventilation and gas exchange, and spectroscopic indices will be evaluated to test gas exchange dynamics with high temporal resolution. The conventional 1H MRI scans will include a free-breathing ultra-short echo time (UTE) scan that provides images similar to that of a CT scan.

ELIGIBILITY:
Inclusion Criteria:

Patients with known Pulmonary Hypertension on treatment with inhaled prostacyclin (iTRE) that are followed in the Duke Pulmonary Vascular Disease Clinic. Inclusion criteria includes: Group 1 PH (mPAP ≥ 25 mmHg, PCWP ≤ 15 mmHg in the absence of significant concomitant left heart disease or lung disease), out-of-proportion Group 3 PH (mPAP ≥ 25 mmHg, PCWP ≤ 15 mmHg with PVR ≥ 5 WU and evidence of right heart failure in the setting of lung disease), maintenance on a stable, well-tolerated treatment dose of iTRE (ideally ≥ 8 breaths QID)

Exclusion criteria:

Pregnant women were excluded from this study. Women of childbearing potential must have a negative urine pregnancy test in order to participate in this study.

Definition of Women of CBP: The median age of menopause in the US, defined as 12 months of amenorrhea, is 51 years; by age 48, approximately 15% of women will be postmenopausal, while virtually 100% will be post-menopausal by age 53. Women are considered past the age of "child-bearing potential" if

* they are greater than 55 years of age, OR
* they are at least 50 years of age AND o have not menstruated for at least 12 months, OR
* have a documented Follicule Stimulating Hormone (FSH) level of greater than 40 mIU/mL.
* they are at least 45 years of age AND o have not menstruated for at least 18 months, OR
* have a documented Follicule Stimulating Hormone (FSH) level of greater than 40 mIU/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Rajagopal, MD, PhD, Principal Investigator — Duke University; Bastiann Driehays, PhD, Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulmonary Hypertension Patients on Inhaled Prostacyclin: 11 subjects will Pulmonary Hypertension on a stable dose of Inhaled Prostacyclin for treatment of PH.
  Hyperpolarized 129Xenon gas: Hyperpolarized 129Xenon gas XeMRI scans will provide 3D images of ventilation and gas exchange pre, post, and 2-4 hours post inhaled prostacyclin treatment. Subjects will inhale HP 129Xe from the dose delivery bags with each scan and then move into the scanner and undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will undergo several MRI scans after inhalation of HPXe. This will occur as three scans at the three different time points (pre, post, and 2-4 hours post) of inhaled prostacyclin treatment.
Period: Overall Study
Arm/Group | Pulmonary Hypertension Patients on Inhaled Prostacyclin
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Same as participant flow information
Groups:
- Pulmonary Hypertension Patients Treated With Inhaled Treprostinil (iTRE): Patients with known PH on treatment with iTRE that are followed in the Duke Pulmonary Vascular Disease Clinic.
Arm/Group | Pulmonary Hypertension Patients Treated With Inhaled Treprostinil (iTRE)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [63 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Abnormal RBC Percentage
Description: Percent change in pulmonary gas exchange (percent change in abnormal RBC percentage - calculated as: 100*(value at 3 hours - value at baseline)/value at baseline) in patients with PH treated with inhaled prostacyclin.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pulmonary Hypertension Patients on Inhaled Prostacyclin
Number analyzed (Participants) | 11
percent change | -17.7 (24.4)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Pulmonary Hypertension Patients on Inhaled Prostacyclin
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT03367312/Prot_SAP_ICF_000.pdf